CLINICAL TRIAL: NCT00773721
Title: Assessment of Bioburden in a New Mask Seal Material
Brief Title: Foam Mask - Assessment of Bioburden in a New Mask Seal Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA131008
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Volunteers who are currently using CPAP treatment will trial a new mask system for up to five weeks
  Interventions: Device: CPAP mask

INTERVENTIONS:
Device: CPAP mask — Current CPAP masks are mainly silicone elastomers, which though well understood and accepted, are often uncomfortable.
  Test Units: The test unit is a foam seal component which directly replaces the patients existing silicone mask cushion, and is fitted to the patients existing mask frame.
  Subjects will wear the test unit mask, instead of their current CPAP mask, each night whilst sleeping.

SUMMARY:
Obstructive sleep apnoea (OSA) is characterised by a partial or complete collapse of the upper airway during sleep. The treatment of choice for OSA is Continuous Positive Airway Pressure (CPAP). CPAP acts as a positive airway splint, delivering a fixed positive airway pressure to the upper airway via a tube and mask. Compliance, however, to therapy requires that the mask is suitably comfortable so as not to disturb sleep.

A key contributor to comfort is the seal component of the mask system. Current mask seals are mainly silicone elastomers, which though well understood and accepted, are often uncomfortable. It is proposed to replace the solid elastomer with a soft polymer foam.

The foam is highly porous, and has open cells at its surface. It is therefore more likely to accumulate biological material with repeated use. The current (silicone) material does not present any problematic bioburden issues. Therefore it is important to investigate whether the foam will present bioburden problems to patients, within specified usage parameters.

The aims of this study therefore are:

1. to observe the rate of bacterial accumulation on foam mask seal material (polyether polyurethane,)
2. to determine the replacement interval for a foam mask seal, and
3. assess the comfort and function of a foam mask seal.

DETAILED DESCRIPTION:
Test Units: The test unit is a foam seal component which directly replaces the patients existing silicone mask cushion, and is fitted to the patients existing mask frame.

Subjects will wear the test unit mask, instead of the current CPAP mask, each night whilst sleeping. Upon waking, subjects will remove the test unit mask and place it with the skin contact side uppermost on a flat surface adjacent to their bed (e.g. a bedside table). Test unit masks should not be covered, and are to remain exposed to the bedroom environment for the rest of the day. The cycle repeats for up to 35 days (5 weeks).

If necessary, the test can be terminated before this time.

A control group of 2 subjects will wash their test unit mask with only hot water every day for the 5 weeks. Another 4 subjects will have the foam of their test unit mask replaced during the 5 weeks of the trial. Two subjects will have the foam changed after 2 weeks and the other 2 subjects after 4 weeks. This will allow estimations of bioburden after 1,2,3,4 and 5 weeks of use.

The foam samples are to be sealed in the supplied sterile container. The sealed container will be delivered as soon as possible to the project administrator. The project administrator will appropriately collect, record, store, and dispatch the sealed samples for microbiological analysis.

Microbial analysis will determine the number of colony forming units, and species present in each test unit upon test termination.

Skin Reactions:

Participants will be asked to report any skin reaction they experience under the test unit. Subjects will keep a bi-weekly record of any skin redness, irritation, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18+
* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients being treated for OSA with CPAP for >6 months
* Patients using ResMed Masks

Exclusion Criteria:

* • Known to have any pre-existing dermatological condition

  * Has been treated with antibiotics in the previous month
  * Any condition which, in the opinion of the investigator, would make the subject unsuitable or unsafe for enrolment, or could interfere with the subject participating in and completing the protocol.
  * Patients currently using ResMed masks: Swift, Activa, or Liberty.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Measurement of bacterial accumulation in the new material. | up to 35 days (5 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, PhD, Principal Investigator — ResMed/ The University of New South Wales
Locations (1):
- Resmed Centre for Healthy Sleep, Sydney, New South Wales, Australia